CLINICAL TRIAL: NCT06431568
Title: Effect of Prophylactic IV Ondansetron Prior Spinal Anaesthesia in Caesarean Section on Bradycardia and Hypotension (Observational Study)
Brief Title: Ondansetron Prior Spinal Anaesthesia
Acronym: Ondansetron
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Collaborators: Kuwait Institute for Medical Specialization (Other Government)
Responsible Party: Principal Investigator, Abdelrady S Ibrahim, MD, Professor of Anesthesia and ICU, Assiut University
Other Study IDs: IRB0000871252; Kuwait MOH (Other: Maternity Hospital)
Record Dates: First submitted 2024-05-22; First posted 2024-05-28 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-05

CONDITIONS: Cesarean Section
Keywords: Spinal anesthesia, Cesarean section, Ondansetron

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Intravenous Ondansetron for patients undergoing Cesarean section under spinal Anesthesia: Pregnant patients undergoing elective caesarean section with no co-morbidities will receive intravenous ondansetron

SUMMARY:
Since Ondansetron is commonly used during cesarean deliveries to treat nausea and vomiting, this study will observe the correlation between ondansetron administration and effect on hemodynamics in order to confirm that the use of Ondansetron can reduce incidence of hypotension and bradycardia associated with spinal in cesarean section, and to identify the optimal timing and dose for administration.

DETAILED DESCRIPTION:
Hypothesis:

Administration of ondansetron prior to spinal anesthesia can attenuate hypotension and bradycardia.

Aim:

Since Ondansetron is commonly used during cesarean deliveries to treat nausea and vomiting, this study will observe the correlation between ondansetron administration and effect on hemodynamics in order to confirm that the use of Ondansetron can reduce incidence of hypotension and bradycardia associated with spinal in cesarean section, and to identify the optimal timing and dose for administration.

Objectives:

* Primary outcome: incidence of hypotension after spinal anaesthesia in the patients who received Ondansetron and those who did not
* Secondary outcome : use of vasopressors , bradycardia , timing of administration of Ondansetron wether it is more or less than five minutes prior to the administration of anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant patients undergoing elective caesarean section

Exclusion Criteria:

* Preeclampsia
* Eclampsia
* Hypertension
* Diabetes

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Pregnant patients undergoing elective cesarean section with no co-morbidities before or during pregnancy period
Study Population: Pregnant patients undergoing elective caesarean section with no co-morbidities before or during pregnancy period, e.g. HTN, DM, PET or Eclampsia, will be recruited. Attempt will be made to include all eligible participants
Sampling Method: Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-03-02 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Blood Pressure | one hour
  incidence of hypotension after spinal anaesthesia in the patients who received Ondansetron

SECONDARY OUTCOMES:
Heart rate | One hour
  Incidence of bradycardia after ondansetron
Vasopressor | One hour
  Incidence of use of ephedrine or phenylpherine

CONTACTS AND LOCATIONS:
Overall Officials: Abdelrady S Ibrahim, .M.D., Principal Investigator — Assiut University Faculty Of Medicine
Locations (1):
- Assiut university faculty of medicine, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Hofhuizen C, Lemson J, Snoeck M, Scheffer GJ. Spinal anesthesia-induced hypotension is caused by a decrease in stroke volume in elderly patients. Local Reg Anesth. 2019 Mar 4;12:19-26. doi: 10.2147/LRA.S193925. eCollection 2019. PMID 30881108